CLINICAL TRIAL: NCT04545437
Title: The Short and Long-term Cardiovascular Consequences of Critical Illness: The C3 Study
Acronym: C3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID14762; Oxford Rec C (Other: 20/SC/0105); Confidentiality Advisory Group (Other: 20/CAG/0038)
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Critical Illness; Myocardial Infarction; Stroke; Atrium; Fibrillation; Atrial Flutter
MeSH Terms: conditions — Critical Illness; Myocardial Infarction; Stroke; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU: Patients treated on a general adult intensive care unit
  Interventions: Other: Admission to ICU

INTERVENTIONS:
Other: Admission to ICU — Exposure is admission to an Intensive Care Unit

SUMMARY:
The aim this study will be to find out which patients are at risk of heart attacks/strokes up to several years after discharge from an ICU. This study will also investigate whether treatments and events occurring in ICU contribute to this risk.

DETAILED DESCRIPTION:
Undertake a retrospective observational cohort study of patients admitted to intensive care units between 2006 and 2023.

Study Participants: Adult patients admitted to a general adult intensive care unit at one or more of the study sites between 2006 and 1st of August 2023.

Objectives:

To determine the short and long-term cardiovascular consequences of critical illness and identify in-ICU factors that affect them.

To identify the risk factors for new-onset atrial fibrillation/flutter occurring during critical illness.

To study the association between poor cardiovascular function during critical illness and long-term cardiovascular disease.

This study will provide new knowledge about the associations between baseline cardiovascular risk, the disease resulting in ICU admission and therapies / events on ICU with subsequent major adverse cardiac events (MACE), to allow the ongoing risk of these events to be determined. If clinicans can idetnify who is at risk, then risk factors can potentially be modified .

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or above.
* Admitted to an intensive care unit at a study site from 2006 onwards

Exclusion Criteria:

* Patients that have informed their participating site that they do not wish their electronic records would be used for future research
* Patients who inform us directly that they don't wish their records used in this research study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients admitted to a general adult intensive care unit at one or more of the study sites between 2006 and 1st of August 2023.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
Major adverse cardiovascular and vascular events | 5 years
Arrhythmia | 5 years

SECONDARY OUTCOMES:
Hospital re-admission | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Watkinson, Study Director — University of Oxford
Locations (3):
- United Kingdom (3):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - Oxford University Hospitals, Oxford, Oxfordshire
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publically available due to privacy and legal implications. Secondary analysis of the study will be considered on a case by case basis.

REFERENCES:
- See also: Critical Care Research Group main website — https://www.ndcn.ox.ac.uk/research/critical-care-research-group-kadoorie-centre